CLINICAL TRIAL: NCT05669430
Title: An Open-Label Phase 1/2A Study of GV20-0251 Monotherapy and GV20-0251 in Combination With Pembrolizumab in Participants With Advanced and/or Refractory Solid Tumor Malignancies
Brief Title: A Study of GV20-0251 Monotherapy and GV20-0251 in Combination With Pembrolizumab in Participants With Solid Tumor Malignancies
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: GV20 Therapeutics (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GV20-0251-100; GV20-0251-100 (Other: GV20 Therapeutics); MK-3475-F77 (Other: Merck); KEYNOTE-F77 (Other: Merck)
Record Dates: First submitted 2022-12-12; First posted 2022-12-30 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Solid Tumor, Adult; Refractory Cancer; Endometrial Carcinoma (EC); Squamous Head and Neck Carcinoma; pMMR/MSS Adenocarcinoma of the Colon or Rectum; Cutaneous Melanoma; Non-Small Cell Lung Cancer
Keywords: GV20-0251
MeSH Terms: conditions — Neoplasms; Endometrial Neoplasms; Melanoma; Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part A - Dose Escalation in up to 7 dose levels (Experimental): A 3+3 dose escalation scheme will be used to evaluate the safety and tolerability of GV20-0251, and to establish the maximum tolerated dose (MTD) or the preliminary recommended Phase 2 dose (RP2D).
  Interventions: Biological: GV20-0251
- Part B - Multiple Expansion Cohorts in up to 4 tumor indications (Experimental): The Bayesian optimal design for Phase II (BOP2) will be utilized to further characterize the anti-tumor activities, safety, tolerability, pharmacokinetics, and pharmacodynamics of GV20-0251 at the preliminary RP2D in up to 4 expansion cohorts involving eligible participants.
  Interventions: Biological: GV20-0251
- Part C - GV20-0251 in Combination with Pembrolizumab Dose Escalation in 2-4 dose levels (Experimental): The Bayesian optimal interval (BOIN) design will be employed to evaluate the safety and tolerability of GV20-0251 in combination with pembrolizumab, and to determine the MTD or the preliminary RP2D of this combination in selected tumor indications.
  Interventions: Biological: GV20-0251 and Pembrolizumab [KEYTRUDA®]
- Part D - GV20-0251 in Combination with Pembrolizumab Dose Expansion in up to 5 indications (Experimental): The BOP2 will be applied to further characterize the anti-tumor activities, safety, tolerability, pharmacokinetics, and pharmacodynamics of GV20-0251 in combination with pembrolizumab at the preliminary RP2D in up to 5 expansion cohorts involving eligible participants.
  Interventions: Biological: GV20-0251 and Pembrolizumab [KEYTRUDA®]

INTERVENTIONS:
Biological: GV20-0251 — Increasing doses of GV20-0251 administered by intravenous (IV) infusion once or twice every 3 weeks as monotherapy.
  Arms: Part A - Dose Escalation in up to 7 dose levels
Biological: GV20-0251 — GV20-0251 preliminary RP2D administered by IV infusion as monotherapy.
  Arms: Part B - Multiple Expansion Cohorts in up to 4 tumor indications
Biological: GV20-0251 and Pembrolizumab [KEYTRUDA®] — GV20-0251 administered by IV infusion at 10 mg/kg once every 3 weeks or at increasing doses up to the preliminary RP2D determined in Part A. 200 mg pembrolizumab administered by IV infusion once every 3 weeks.
  Other Names: MK-3475
  Arms: Part C - GV20-0251 in Combination with Pembrolizumab Dose Escalation in 2-4 dose levels
Biological: GV20-0251 and Pembrolizumab [KEYTRUDA®] — GV20-0251 administered by IV infusion at preliminary RP2D from Part C. 200 mg pembrolizumab administered by IV infusion once every 3 weeks.
  Other Names: MK-3475
  Arms: Part D - GV20-0251 in Combination with Pembrolizumab Dose Expansion in up to 5 indications

SUMMARY:
This is a Phase 1/2A study of GV20-0251 being developed for the treatment of participants with advanced solid tumors, who are refractory to approved therapies or other standard of care.

DETAILED DESCRIPTION:
This is a Phase 1/2A non-randomized, open label, multi-center study to be conducted in four parts (Parts A, B, C and D).

In Part A, a 3+3 dose escalation scheme will be used to evaluate the safety and tolerability of GV20-0251, and to establish the maximum tolerated dose (MTD) or the preliminary recommended Phase 2 dose (RP2D).

In Part B, the Bayesian optimal design for Phase II (BOP2) will be utilized to further characterize the anti-tumor activities, safety, tolerability, pharmacokinetics, and pharmacodynamics of GV20-0251 at the preliminary RP2D across multiple expansion cohorts involving eligible participants.

In Part C, the Bayesian optimal interval (BOIN) design will be employed to evaluate the safety and tolerability of GV20-0251 in combination with Pembrolizumab, and to determine the MTD or the preliminary RP2D of this combination.

In Part D, BOP2 will be applied to further characterize the anti-tumor activities, safety, tolerability, pharmacokinetics, and pharmacodynamics of GV20-0251 in combination with Pembrolizumab at the preliminary RP2D across multiple expansion cohorts involving eligible participants.

ELIGIBILITY:
Inclusion Criteria:

* Participants ≥18 years of age
* Previously treated, histologically-confirmed advanced solid malignancy with progressive disease requiring therapy
* Refractory or intolerant to standard therapy(ies)
* Must have received, be not eligible or decline standard of care therapy
* Participants must have measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST version 1.1)
* For participants who have received prior treatment with a checkpoint inhibitor there must be documented disease progression
* ECOG performance status of 0 or 1
* Life expectancy of ≥ 12 weeks in Parts A and C and ≥ 24 weeks in Parts B and D
* Participants must be willing to provide fresh tumor biopsy (core biopsy) both pre-treatment (Parts A, B, C and D) and on-treatment (Parts A and B), if clinically feasible
* Disease-free of active second/secondary or prior malignancies for ≥ 2 years
* Laboratory test results within the required parameters
* Women of child bearing potential (WOCBP) and men must agree to use adequate contraception
* Parts B, C and D may include the following tumor types:

  * Endometrial carcinoma
  * Squamous head and neck carcinoma
  * Cutaneous melanoma
  * Non-small cell lung cancer
  * Proficient MMR (pMMR)/MSS adenocarcinoma of the colon or rectum (Parts C and D only)

Parts A, B, C and D Exclusion Criteria:

* Participant with acute leukemia or CLL (Parts A and B only)
* Participant with heart disease or unstable arrhythmia
* Active, uncontrolled bacterial, viral, or fungal infections requiring systemic therapy
* Participant has active autoimmune disease or other medical conditions requiring chronic systemic steroid or immunosuppressive therapy
* History of major organ transplant
* History of a bone marrow transplant
* Symptomatic central nervous system (CNS) malignancy or metastasis
* Serious nonmalignant disease
* Pregnant or nursing women
* Treatment with PD-1 and equivalent immune modulators or major surgery prior to the first dose of study medication
* Participants who are currently receiving any other investigational agent or have received an investigational agent within 4 weeks prior to the first dose of study medication
* Treatment with any anticancer treatments with 2-weeks prior to the first dose of study medication
* Radiation for symptomatic lesions must have been completed prior to the first dose of study medication
* Participants with liver metastases unless approved by the Sponsor
* Any history of an immune related ≥ Grade 3 AE attributed to prior cancer immunotherapy
* Has a known additional malignancy that is progressing or has required active treatment within the past 2 years from C1D1
* Has received radiation therapy to the lung that is higher than 30 Gy within 6 months prior to C1D1 for NSCLC (Parts C and D only)
* Has a known additional malignancy that is progressing or has required active treatment within the past 2 years from C1D1 (Parts C and D only)
* Has severe hypersensitivity ( ≥ Grade 3) to Pembrolizumab and/or any of its excipients (Parts C and D only)
* Has a history of (non-infectious) pneumonitis / interstitial lung disease that required steroids or has current pneumonitis / interstitial lung disease (Parts C and D only)
* Has a condition, therapy, laboratory abnormality, or circumstance that could confound study results or interfere with full participation, making it unsuitable for the participant, as determined by the treating Investigator (Parts C and D only)
* Active substance abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 365 (Estimated)
Dates: Start 2023-03-23 (Actual); Primary Completion 2026-12-15 (Estimated); Study Completion 2027-09-05 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate ORR per RECIST version 1.1 (Parts B and D) | 12 months
  ORR
Percentage of Participants With Adverse Events (Parts A and C) | 12 months

SECONDARY OUTCOMES:
Overall Survival (Parts B and D) | 24 months
  OS
Additional safety and tolerability | 24 months
  TEAEs per NCI CTCAE version 5.0
Cmax of GV20-0251 | 12 months
  Maximum concentration
Tmax of GV20-0251 | 12 months
  Time to peak drug concentration
T1/2 | 12 months
  Terminal half-life of GV20-0251
AUC | 12 months
  Area under the curve
ADAs | 12 months
  Specification and quantification of anti-drug antibodies
nADAs | 12 months
  Neutralizing anti-drug antibodies
DCR | 24 months
  Disease Control Rate is the percentage of participants with stable disease, complete response or partial response among all response evaluable participants
DoR | 24 months
  Duration of Response is the time from first CR/PR to the date of PD or death.
PFS | 24 months
  Progression Free Survival is the duration from the first dose to PD/death
ORR (Parts A and C) | 24 months
  Percentage of participants with complete response or partial response among all response evaluable participants

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - The Angeles Clinic and Research Institute, Los Angeles, California
  - HealthONE Clinic Services Oncology - Hematology, LLC d/b/a Sarah Cannon Research Institute at HealthONE, Denver, Colorado
  - Yale University, New Haven, Connecticut
  - Florida Cancer Specialists & Research Institute, LLC, Fort Myers, Florida
  - Community Health Network, Inc., Indianapolis, Indiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Barbara Ann Karmanos Cancer Hospital dba Karmanos Cancer Center, Detroit, Michigan
  - NYU Langone Health, New York, New York
  - Oregon Health & Science University, Portland, Oregon
  - Verdi Oncology Tennessee, Scri Oncology Partners, Nashville, Tennessee
  - Oncology Consultants, P.A., Houston, Texas
  - The University of Texas M. D. Anderson Cancer Center, Houston, Texas
  - Virginia Cancer Specialists, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li Y, Wu X, Sheng C, Liu H, Liu H, Tang Y, Liu C, Ding Q, Xie B, Xiao X, Zheng R, Yu Q, Guo Z, Ma J, Wang J, Gao J, Tian M, Wang W, Zhou J, Jiang L, Gu M, Shi S, Paull M, Yang G, Yang W, Landau S, Bao X, Hu X, Liu XS, Xiao T. IGSF8 is an innate immune checkpoint and cancer immunotherapy target. Cell. 2024 May 23;187(11):2703-2716.e23. doi: 10.1016/j.cell.2024.03.039. Epub 2024 Apr 23. PMID 38657602
- [Result] Wentzel, K., Peguero, J., Kummar, S., Lorusso, P., Mehnert, J. M., Spira, A. I., Naing, A., Hamid, O., Mehmi, I., Benhadji, K., Alland, L., Hu, X., Xiao, H., Bao, X., Chen, J., Gong, Y., Liu, X. S. ESMO 2024
- See also: IGSF8 is an innate immune checkpoint and cancer immunotherapy target — https://doi.org/10.1016/j.cell.2024.03.039
- See also: A phase I/II, open-label study of the novel checkpoint IGSF8 inhibitor GV20-0251 in patients with advanced solid tumors — https://doi.org/10.1016/j.annonc.2024.08.1059